CLINICAL TRIAL: NCT05741515
Title: Feasibility of a Home-Based Vestibular Balance Therapy Intervention for Children With Vestibular Hypofunction
Brief Title: Vestibular Balance Therapy Intervention for Children
Acronym: VBT-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Foundation for Physical Therapy Research (Other)
Responsible Party: Principal Investigator, Jennifer Braswell Christy, Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300010569
Record Dates: First submitted 2023-01-25; First posted 2023-02-23 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Vestibulocochlear Nerve Diseases; Vestibular Disorder; Bilateral Vestibular Loss
Keywords: pediatric; vestibular rehabilitation; dynamic visual acuity; postural control; feasibility
MeSH Terms: conditions — Vestibulocochlear Nerve Diseases; Vestibular Diseases; Bilateral Vestibulopathy

STUDY DESIGN:
Intervention Model Description: prospective single arm feasibility clinical trial. We will also enroll 3 children in a control intervention group, but these will be children without the condition, to determine the feasibility of the control intervention.
Who Masked: Outcomes Assessor
Masking Description: The clinicians doing the functional outcome measures (FGA, DVA, SOT) will not know the result of the vestibular function tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VBP Intervention Group (Experimental): Children coded as abnormal on functional tests (FT) (n=12) will participate in an 8-week 5X/week home-based VBT program. At the initial visit (T0), the PI will instruct the participants (caregiver and child) in the program and provide all materials. The exercises will be led by the caregiver, with weekly in person checks by the PI to progress and provide coaching. The child/caregiver will complete a daily log to report activities and level of enjoyment. VBT will be done 5 days/week and will include 4 key categories of exercises, each lasting 5 minutes (20 minutes total of exercise per day). The 4 categories, explained below, include: 1) Times 1 (X1) Viewing, 2) Gaze Shifting, 3) Static Balance, 4) Dynamic Balance. The proposed VBT home program will include 10 minutes of gaze stabilization exercises, and 10 minutes of balance training.
  Interventions: Other: Vestibular Balance Therapy
- Sham Intervention (Sham Comparator): Sham Intervention (not to be compared to intervention - for feasibility only):
  Aim 1 is to establish the feasibility of a control intervention to be used in future studies. Therefore, 3 participants who score above the set criterion for the Functional Tests (FT) (i.e., they do not need VBT) will participate in an 8-week sham intervention. At T0, the PI will instruct the participants to do the sham intervention, led by the caregiver with weekly checks to control for attention bias. The sham intervention will be done for 20 minutes per day and will consist of 10 minutes of focused reading a book of the child's choice and 10 minutes of active play. The child and caregiver will complete a daily activity log documenting the activity and level of enjoyment.
  Interventions: Other: Sham Intervention

INTERVENTIONS:
Other: Vestibular Balance Therapy — see intervention arm description
  Other Names: Vestibular Rehabilitation
  Arms: VBP Intervention Group
Other: Sham Intervention — see sham intervention arm description
  Arms: Sham Intervention

SUMMARY:
The goal of this within groups clinical trial is to determine the feasibility of a home-based vestibular balance therapy program for children with vestibular hypofunction. The main questions to be answered are: 1) what is the intervention's feasibility and 2) what is the intervention's preliminary impact on function? Participants will receive a comprehensive battery of vestibular function and balance tests, then an 8-week home-based intervention to be done 5 times/week with weekly checks from the physical therapist. Data will be used to design a larger clinical trial with a comparison group.

DETAILED DESCRIPTION:
Approximately 60-75% of children with severe/profound sensorineural hearing loss (SNHL) also have vestibular hypofunction (VH), resulting in delayed gross motor development, poor postural control, and gaze instability. Although clinical practice guidelines provide recommendations for adults with VH, no statements exist for children due to a paucity of high- level studies. The long-term objective of this proposal is to assess feasibility of a home-based vestibular balance therapy (VBT) program for children so that a larger well-powered controlled study can be designed. The specific aims are to assess the intervention's feasibility (Aim 1), estimate its preliminary impact on functional outcomes (Aim 2), and assess participant engagement (secondary Aim). To accomplish this, we will use a prospective single arm feasibility design. We will enroll 15 children with SNHL, aged 4-17 years; 12 with confirmed VH for the VBT, and 3 with normal vestibular function to test the sham intervention. All children will be tested on the functional outcomes: computerized dynamic visual acuity, modified functional gait assessment, and sensory organization test at baseline, 4, and 8 weeks. A physical therapist (PT) will train children/caregivers in the 8-week structured VBT home program consisting of 4 categories of exercises (Times 1 viewing, gaze shifting, static and dynamic balance) done 5 times/week, 5 minutes/exercise. The PT will meet weekly with the child/caregiver in person to systematically progress the exercises. The children in the sham intervention (10 minutes of reading, 10 minutes of play) will also receive weekly meetings with the PT to control for attention bias. To assess Aim 1 (Feasibility) metrics will include process (e.g., recruitment rates), resources (e.g., communication needs), management (e.g., data collection/entry), experience (e.g., barriers). To assess Aim 2 (impact) we will analyze within group changes and effect sizes to design the larger study.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of severe to profound SNHL
* age 4-17 years
* caregiver/child verbal willingness to commit to the home vestibular balance therapy or sham intervention
* vision screening/testing within 1 year or willingness to get a vision test.

Exclusion Criteria:

* neurologic condition other than SNHL
* inability to read at a kindergarten level or identify pictures
* currently receiving vestibular therapy
* uncorrected vision problems unrelated to a vestibular deficit

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Change in Computerized Dynamic Visual Acuity at 4 and 8 weeks | Baseline (pre), 4 weeks (mid), 8 weeks (post)
  Difference in visual acuity with the head stationary versus moving
Change in Functional Gait Assessment at 4 and 8 weeks | Baseline (pre), 4 weeks (mid), 8 weeks (post)
  A standardized test of dynamic balance
Change in Sensory Organization Test at 4 and 8 weeks | Baseline (pre), 4 weeks (mid), 8 weeks (post)
  A standardized test of static postural control

SECONDARY OUTCOMES:
Process Feasibility (Recruitment Rates) | through study completion at 2 years
  % of individuals who follow through with enrollment procedures
Process Feasibility (Refusal Rate Frequency) | through study completion at 2 years
  Frequency of refusal to participate in the study
Process Feasibility (Attrition Rates) | through study period at 2 years
  % of attrition
Process Feasibility (Retention Rates) | through study period at 2 years
  % of retention
Process Feasibility (Completion Rates) | through study period at 2 years
  % of participants who complete 80% of intervention sessions
Management Feasibility (training) | through year 1
  time in minutes to train data collectors
Management Feasibility (data entry) | through year 1
  time in minutes for data entry
Participant Experience Feasibility (Strategies) | through study period at 2 years
  participant strategies that helped them with participation in the study (interview)
Participant Experience Feasibility (Enjoyment) | through the study period at 2 years
  Enjoyment level for each participant (ordinal scale of 0=no enjoyment to 10=extreme enjoyment)
Participant Experience Feasibility (Testing Difficulty) | baseline only - initial testing session
  Participants will rate the level of difficulty of the initial testing session (0=not difficult to 10=extreme difficulty)
Participant Experience Feasibility (Intervention Difficulty) | once, at each participant's final testing session (8 weeks)
  Participants will rate the level of difficulty of the overall intervention (0=not difficult to 10=extreme difficulty)
Resource Feasibility (frequency) | through study period at 2 years
  Frequency of communication with participants
Resource Feasibility (time) | through study period at 2 years
  Total time in minutes to communicate with participants

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer B Christy, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI plans to share the data via typical methods such as manuscripts and professional conferences.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be shared after study completion and following analysis. The PI may choose to share preliminary data at a conference.

REFERENCES:
- [Background] Christy JB, Payne J, Azuero A, Formby C. Reliability and diagnostic accuracy of clinical tests of vestibular function for children. Pediatr Phys Ther. 2014 Summer;26(2):180-9. doi: 10.1097/PEP.0000000000000039. PMID 24675116
- [Background] Rine RM, Braswell J. A clinical test of dynamic visual acuity for children. Int J Pediatr Otorhinolaryngol. 2003 Nov;67(11):1195-201. doi: 10.1016/j.ijporl.2003.07.004. PMID 14597370
- [Background] Rine RM, Braswell J, Fisher D, Joyce K, Kalar K, Shaffer M. Improvement of motor development and postural control following intervention in children with sensorineural hearing loss and vestibular impairment. Int J Pediatr Otorhinolaryngol. 2004 Sep;68(9):1141-8. doi: 10.1016/j.ijporl.2004.04.007. PMID 15302144
- [Background] Braswell J, Rine RM. Preliminary evidence of improved gaze stability following exercise in two children with vestibular hypofunction. Int J Pediatr Otorhinolaryngol. 2006 Nov;70(11):1967-73. doi: 10.1016/j.ijporl.2006.06.010. Epub 2006 Oct 4. PMID 17023057